CLINICAL TRIAL: NCT06770400
Title: Optimizing Bedroom Temperature to Improve Sleep in Older Adults
Brief Title: Sleep Improvement Via Environmental Smart Temperature Adjustments
Acronym: SIESTA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Amir Baniassadi, Principal Investigator, Hebrew SeniorLife
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Sleep and Temperature Study
Record Dates: First submitted 2024-09-25; First posted 2025-01-13 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Sleep; Environmental Exposure; Environmental Sleep Disorder
Keywords: Temperature; Sleep; Older adults
MeSH Terms: conditions — Dyssomnias | interventions — Sleep

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): After the initial monitoring, the bedroom temperature for the experimental group will be set to what is deemed optimal for their sleep. Participants will always have the option of overriding our prescribed temperature.
  Interventions: Other: Temperature Optimized for Sleep
- Control (Experimental): After the initial monitoring, the control group will control their own bedroom temperature.
  Interventions: Other: Participant's Preferred Temperature

INTERVENTIONS:
Other: Temperature Optimized for Sleep — Using the cloud-controlled thermostat, we will prescribed bedroom temperature based on the observed relationship between the individual's sleep quality and the temperature of their bedroom.
  Arms: Intervention
Other: Participant's Preferred Temperature — Temperature is set by the individual based on their own habits and preference.
  Arms: Control

SUMMARY:
Nearly 50% of older adults complain of poor habitual sleep, and in many cases the underlying reason remains undiagnosed or unknown. Meanwhile, observational data suggest that bedroom temperature significantly influences sleep quality in community-dwelling older adults, including those without financial constraints that limit the use of heating and cooling. These individuals often struggle to maintain an optimal bedroom temperature, either due to impaired motor function and cognitive abilities, and/or a lack of awareness about how temperature affects their sleep. Therefore, for a non-trivial portion of older adults, optimizing the bedroom temperature presents an exciting and untapped opportunity to improve sleep without substantial cost, burden, and side effects. The intervention, biologically adaptive control of bedroom temperature, uses wearable health trackers (e.g., a Garmin watch) and smart thermostats to automate and personalize bedroom temperature control, tailoring it to each person's unique physiology and context. Initially, individuals will be monitored in their home to determine each person's specific temperature range that promotes sleep quality, as measured by the wearable device. After the initial monitoring, the smart thermostat will maintain bedroom temperature within the optimal range for sleep for as long as the individual uses the intervention.

The primary purpose of this project is to test the feasibility of biologically adaptive control of bedroom temperature as an intervention to improve sleep in older adults and gather preliminary data to facilitate sample size calculations for a definitive trial. 20 Older adults, aged 65 and above, will be enrolled and their bedrooms bedrooms will be equipped with smart thermostats. The first aim focuses on assessing the feasibility of the intervention. This includes evaluating participant recruitment and retention, the acceptability of temperature adjustments (tracked through the number of temperature overrides by participants), and the self-reported likelihood of future use. The second aim involves analyzing the mean and variance of sleep outcomes during observation and intervention phases (separately for each group), examining the degree to which they vary with temperature variations and behavioral adaptations.

DETAILED DESCRIPTION:
Background and Rationale for the Research

Lab-based studies have shown that ambient temperature significantly affects sleep outcomes, such as sleep efficiency, which in turn influences cognitive function, mental health, stress, physical activity, cardiovascular health, and morning glucose levels. Investigator's recent research confirms that bedroom temperature impacts sleep quality even in home settings where individuals can control their environment. In a study monitoring 50 community-dwelling older adults over 18 months, over 11,000 person-nights of sleep data were gathered, revealing that small deviations from the optimal bedroom temperature range can significantly disrupt sleep quality, similar to the effects of chronic pain or late-night alcohol consumption. Importantly, the ideal sleep temperature varies by individual, and while participants had access to heating and cooling systems, many older adults still sleep in uncomfortably hot or cold bedrooms due to limited motor function, cognitive issues, or not realizing how temperature affects their sleep. The proposed intervention automates temperature control, tailoring it to individual sleep needs using wearable devices and smart thermostats. The intervention, which optimizes sleep temperature based on personal monitoring data, offers a cost-effective way to improve the wellbeing of older adults, particularly given its low cost and potential for net energy savings from smart thermostat use.

Hypothesis

Biologically adaptive control of the bedroom temperature as an intervention to improve sleep is feasible in older adult populations.

Aims Aim 1: To test the feasibility of biologically adaptive control of the bedroom temperature as an intervention to improve sleep in older adults; Aim 2: Gather preliminary data to facilitate sample size calculations for a definitive trial.

Study Design

Both aims will be completed by recruiting a cohort of older adults living in Boston. Up to 25 individuals will be enrolled to ensure a minimum of 20 complete the study. Half of the sample will be from subsidized housing, addressing the possible substandard conditions such as poor insulation that contribute to temperature regulation issues. The study will be conducted using a rolling enrollment approach with three data collection campaigns. All aspects of the protocol below (including having two equally sized control and experiment groups in each campaign) will be similar among the data collection campaigns. Participants will wear a Garmin watch to continuously monitor sleep-related metrics, and complete a daily survey to report subjective sleep quality and other relevant factors about the previous night.

Overall Study protocol

Screening and enrollment: Individuals will first undergo a standardized phone screen to determine eligibility. Those meeting the criteria will then receive an in-home visit for further evaluation. If a participant is deemed eligible, they may complete the consenting process and the first visit protocol (see below) during the same visit to streamline the process. Visits 1 and 2 will be scheduled in the month before the start of data collection in each campaign. This timing helps participants get familiar with the protocol and minimizes the gap between baseline assessments and data collection.

First visit: individuals will read and sign an informed consent form approved by the IRB. A medical history questionnaire will be completed and medications, blood pressure, height, weight, and demographic information will be recorded. Montreal Cognitive Assessment (MoCA), Pittsburgh Sleep Quality Index (PSQI), and Center for Epidemiological Studies Depression Scale (CESD-R), will be administered. Finally, study staff will set up the wearable device on their or a study-provided smartphone. Comprehensive training on technology use and written instructions will be provided to each participant and repeated as needed.

Second visit: an HVAC contractor will replace the participant's thermostat with the study-provided Ecobee thermostat and the participant will receive training on how to use the Ecobee thermostat to change the temperature.

Data collection: participants will follow the study protocols for 8 weeks:

1. Keep thermostat connected and plugged-in
2. Wear the Garmin watch continuously and charge it once every 5 days.
3. Respond to a short daily questionnaire
4. Open the wearable app in order to sync data once every 5 days.
5. Completed a follow up phone interview halfway through the protocol (10 minutes).
6. Complete a brief exit interview (10 minutes)

Observation period: The initial two weeks will be purely observational, with participants sleeping at their self-selected temperatures. In the following four weeks, small temperature adjustments will be implemented to observe each participant, at least four times, at temperatures ranging from 1.5°C above to 1.5 °C below their initial range. During this four-week period, each night the thermostat will be remotely adjusted according to a pseudorandom schedule, avoiding a difference of more than 1.5°C between consecutive nights. These artificial exposures to different temperatures are important because the investigators' work so far suggests that the typical ambient temperature range for many may not include the optimal conditions for their sleep. Throughout the study, participants can override the prescribed temperature according to their preferences.

Determining optimal temperature for sleep: Using data from the first six weeks, a model will be developed to link the bedroom temperature to sleep in each subject. The input to this model will be 6 weeks' worth of data from each subject. Using this model, the optimal temperature range for each participant will be determined.

Experiment: At the beginning of week seven, participants will be randomly divided into equally sized 'control' and 'experimental' groups. Participants will be blinded to group assignments. During the final two weeks (7 and 8), the bedroom temperature for the experimental group will be maintained within their individual optimal range, as established using the above method, while the control group repeats the purely observational phase, without any remote temperature adjustments.

Exit visit: Participants will be visited at their home to 1) retrieve the Garmin device and Ecobee thermostat, 2) re-install their own thermostat, 3) Complete a brief exit interview about their comfort, perceived improvements in sleep, and their likelihood of adopting the intervention in the future.

Uses of Devices

Garmin watch is a wearable device that is worn on the wrist like a typical watch. Garmin needs to be paired with the participants' smartphone, or the tablet provided by us. Support will be provided per participants' request, or based on the data itself, that may suggest participants are not using the device correctly or the device is not functioning properly.

Cloud-controlled thermostat: A licensed HVAC technician will temporarily replace participants' home thermostat with a controlled Ecobee thermostat. This thermostat will allow the investigators to remotely adjust participants' home ambient temperature. The investigators will adjust the temperature up to once a day based on the protocol above. Importantly, participants will always be able to override the temperature that the investigators selected at any time by simply changing the setting on the thermostat. While the thermostat is digital, in principle, it is like traditional thermostats where a dial on the touch screen can increase or decrease the temperature. At the end of the project, the HVAC technician will retrieve the cloud-controlled thermostat and reinstall the participant's own thermostat.

Daily questionnaires: Participants will complete a daily questionnaire on the LabFront app. Participants will receive daily reminders to complete the questionnaire. Participants may opt to use paper-based versions of these questionnaires.

Informed Consent

Interested individuals will be asked to provide verbal consent to complete initial eligibility screen during a phone conversation with study personnel. Potentially eligible participants will then be scheduled for an in-person screening visit. Potential participants may be emailed or snail-mailed (per request, and according to their preference) a copy of the informed consent for them to review at their own pace prior to the in-person screening. Written informed consent will be obtained by study personnel at the beginning of this in-person screening visit.

All potential participants will be advised of the fact the joining the study is completely voluntary. The entire document should be reviewed with the participant, either having them read it or asking them to follow along as the staff reads it. When the staff is confident that the participant is completely familiar with the document and understands all the aspects of the informed consent form, it should be signed by the participant in the presence of the staff member and should then be signed by the staff member. All consent forms will be double checked to make sure they are properly signed and dated. Copies of completed consent forms will be given to the participant and the original signed document will be kept on file at the Marcus Institute.

ELIGIBILITY:
Inclusion Criteria:

1. At least 65 years old
2. Willing to follow study protocols for the duration of the study
3. Living in the greater Boston metropolitan area
4. Access to stable internet connection within their home
5. Stable medication
6. Ability to speak and read English

Exclusion Criteria:

Exclusion Criteria have been selected to ensure safety and optimize compliance, while minimizing confounds due to overt disease or conditions that may significantly influence study outcomes. The following exclusion criteria will be used to determine eligibility through a phone interview followed by an in-person screening. The exclusion criteria apply to both phases.

1. Stated plans to not live within current place of residence for the duration of the study
2. Inability to properly use the wearable device or complete the daily questionnaire.
3. Self-report of physician-diagnosed sleep apnea or other diagnosed sleep disorders such as restless legs syndrome and chronic insomnia
4. Inability to ambulate without the assistance of others
5. Self- or proxy-report of physician-diagnosed dementia or overt neurological diseases such as Parkinson's Disease, stroke, or Multiple sclerosis
6. Evidence of severe cognitive impairment defined as a Modified Telephone Interview of Cognitive Status (TICS-m) score < 25
7. Self-report of physician-diagnosed type 2 diabetes mellitus.
8. Lack of a thermostat-controlled heating and cooling system to adjust the bedroom temperature. The existing system must be compatible with the thermostat selected in this study (Ecobee)
9. Self-report of any unstable psychiatric illnesses, such as major depressive disorder, schizophrenia, psychosis.
10. Self-report of unstable medical conditions (active cancer, uncontrolled hypertension, unstable heart disease, heart attack within the past 6 months)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency Assessed by Actigraphy | up to 8 weeks
  the ratio of time asleep to time in bed, measured using actigraphy, ranges from 0 (worse outcome) to 100% (better outcome).

SECONDARY OUTCOMES:
Sleep Quality Assessed by a Questionnaire | up to 8 weeks
  sleep subjective quality of sleep, measured using a Single-Item Sleep Quality Scale. The questionnaire instructions direct the respondent to rate the overall quality of sleep whereby the respondent marks an integer score from 0 to 10, according to the following five categories: 0 = terrible, 1-3 = poor, 4-6 = fair, 7-9 = good, and 10 = excellent.
Sleep Duration Assessed by Actigraphy | up to 8 weeks
  in hours, measured using actigraphy, ranges from 0 to 24 hours. (About 8 hours are better outcomes)
Sleep Onset Latency Assessed by Actigraphy | up to 8 weeks
  time to fall asleep, measured using actigraphy, ranges from 0 (better outcome) to 24 hours (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Amir Baniassadi, Principal Investigator — Hebrew SeniorLife
Locations (1):
- Hebrew SeniorLife, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No